CLINICAL TRIAL: NCT07389876
Title: A Multicenter, Real-world Study on Albumin-bound Paclitaxel-based Second-line Treatment Regimens for Locally Advanced or Metastatic Gastric/Gastroesophageal Junction Adenocarcinoma
Brief Title: Albumin-bound Paclitaxel-based Second-line Treatment Regimens for Locally Advanced or Metastatic G/GEJ Adenocarcinoma
Acronym: G/GEJ
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhu, chief physician, Fudan University
Other Study IDs: FDZL-NabPMGC
Record Dates: First submitted 2026-01-26; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer; Second-line Treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Albumin-Bound Paclitaxel; Immune Checkpoint Inhibitors; Angiogenesis Inhibitors; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A (Albumin-bound Paclitaxel Monotherapy Group): Albumin-bound paclitaxel: 112.5 mg/m2, ivgtt, d1, d8, Q3W
  Interventions: Drug: Albumin-bound Paclitaxel
- Group B (Albumin-bound Paclitaxel and Anti-angiogenic Therapy Group): Fruquintinib 4 mg/d, qd po, d1-14, Q3W or Ramucirumab 8 mg/kg d1, 15 Q4W; Albumin-bound paclitaxel: 112.5 mg/m2, ivgtt, d1, d8, Q3W
  Interventions: Drug: Albumin-bound Paclitaxel; Drug: Anti-angiogenic drug
- Group C (Albumin-bound Paclitaxel and Immune Checkpoint Inhibitor Group): Immune checkpoint inhibitor (refer to the drug instructions); Albumin-bound paclitaxel: 112.5 mg/m2, ivgtt, d1, d8, Q3W
  Interventions: Drug: Albumin-bound Paclitaxel; Drug: Immune Checkpoint Inhibitor
- Group D (Albumin-bound Paclitaxel, Immune Checkpoint Inhibitor and Anti-angiogenic Therapy Group): : Fruquintinib 4 mg/d, qd po, d1-14, Q3W or Ramucirumab 8 mg/kg d1, 15 Q4W; Immune checkpoint inhibitor (refer to the drug instructions); Albumin-bound paclitaxel: 112.5 mg/m2, ivgtt, d1, d8, Q3W
  Interventions: Drug: Albumin-bound Paclitaxel; Drug: Immune Checkpoint Inhibitor; Drug: Anti-angiogenic drug
- Group E (Albumin-bound Paclitaxel and Trastuzumab Emtansine Group): Trastuzumab emtansine (first dose 800 mg/m2, subsequent doses 600 mg/m2), ivgtt, Q3W; Albumin-bound paclitaxel: 112.5 mg/m2, ivgtt, d1, d8, Q3W
  Interventions: Drug: Albumin-bound Paclitaxel; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Albumin-bound Paclitaxel — This is a prospective observational study. We observe efficacy and survival of different treatment regimen.
Drug: Immune Checkpoint Inhibitor — Immune Checkpoint Inhibitor
  Groups: Group C (Albumin-bound Paclitaxel and Immune Checkpoint Inhibitor Group); Group D (Albumin-bound Paclitaxel, Immune Checkpoint Inhibitor and Anti-angiogenic Therapy Group)
Drug: Anti-angiogenic drug — Anti-angiogenic drug
  Groups: Group B (Albumin-bound Paclitaxel and Anti-angiogenic Therapy Group); Group D (Albumin-bound Paclitaxel, Immune Checkpoint Inhibitor and Anti-angiogenic Therapy Group)
Drug: Trastuzumab emtansine — Trastuzumab Emtansine
  Groups: Group E (Albumin-bound Paclitaxel and Trastuzumab Emtansine Group)

SUMMARY:
This study is an open-label, multi-cohort real-world research that explores the efficacy and safety of different second-line treatment regimens for gastric/gastroesophageal junction adenocarcinoma that has failed first-line fluoropyrimidine, platinum-based chemotherapy combined with immunotherapy.

DETAILED DESCRIPTION:
Group A (Albumin-bound Paclitaxel Monotherapy Group): Albumin-bound paclitaxel: 112.5 mg/m², intravenous infusion, on days 1 and 8, every 3 weeks.

Group B (Albumin-bound Paclitaxel with Anti-angiogenic Therapy Group): Fruquintinib 4 mg/day, once daily orally, on days 1 to 14, every 3 weeks or Ramucirumab 8 mg/kg on days 1 and 15, every 4 weeks; Albumin-bound paclitaxel: 112.5 mg/m², intravenous infusion, on days 1 and 8, every 3 weeks.

Group C (Albumin-bound Paclitaxel with Immune Checkpoint Inhibitor Group): Immune checkpoint inhibitor (refer to the drug instructions); Albumin-bound paclitaxel: 112.5 mg/m², intravenous infusion, on days 1 and 8, every 3 weeks.

Group D (Albumin-bound Paclitaxel with Immune Checkpoint Inhibitor and Anti-angiogenic Therapy Group): Fruquintinib 4 mg/day, once daily orally, on days 1 to 14, every 3 weeks or Ramucirumab 8 mg/kg on days 1 and 15, every 4 weeks; PD-1 200mg d1, Q3W; Albumin-bound paclitaxel: 112.5 mg/m2, i.v. infusion, on days 1 and 8, every 3 weeks.

Group E (albumin-bound paclitaxel and trastuzumab emtansine group): Trastuzumab emtansine group (initial dose 800 mg/m2, subsequent doses 600-800 mg/m2); Albumin-bound paclitaxel: 112.5 mg/m2, i.v. infusion, on days 1 and 8, every 3 weeks (only patients with Claudin18.2 positive and who did not receive trastuzumab emtansine in the first-line treatment were included).

Treatment continued until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand this study and voluntarily sign the informed consent form;
* Between 18 and 80 years old (inclusive), male or female;
* Patients with unresectable locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma confirmed by pathology or histology;
* ECOG performance status 0-2;
* Known HER2 negative;
* Expected survival ≥ 3 months;
* Patients who have progressed on first-line systemic treatment with fluoropyrimidine-platinum combination and PD-1/PD-L1 monoclonal antibody, or those who have progressed during maintenance treatment; patients with locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma who have progressed within 6 months after the end of perioperative chemotherapy or adjuvant chemotherapy (counting from the end of the combined regimen);
* Have not received taxane-based therapy previously;
* Have at least one measurable lesion (meeting RECIST v1.1 criteria);
* The functions of important organs meet the following requirements (no blood components or cell growth factors are allowed to be used within 14 days before enrollment):

Absolute neutrophil count ≥ 1.5×109/L, white blood cell count ≥ 3.0×109/L; Platelet count ≥ 90×109/L; Hemoglobin ≥ 8g/dL; Total bilirubin (TBIL) ≤ 1.5×ULN; ALT and AST ≤ 2.5×ULN; BUN and creatinine (Cr) ≤ 1.5×ULN (and creatinine clearance (CCr) ≥ 50mL/min); Left ventricular ejection fraction (LVEF) ≥ 50%; Fridericia-corrected QT interval (QTcF) < 470 milliseconds; INR ≤ 1.5×ULN, APTT ≤ 1.5×ULN; Thyroid function: TSH ≤ upper limit of normal (ULN). If abnormal, FT3 and FT4 levels should be examined. If FT3 and FT4 levels are normal, the patient can be enrolled; Premenopausal women and postmenopausal women for less than 1 year must have a negative serum or urine pregnancy test before treatment.

Exclusion Criteria:

* Patients with other malignancies within 5 years before enrollment, except for skin basal cell or squamous cell carcinoma after radical surgery, or cervical carcinoma in situ;
* Patients who have received allogeneic bone marrow transplantation or organ transplantation in the past;
* Patients with severe cardiovascular diseases within 6 months before enrollment, including unstable angina or myocardial infarction;
* Patients allergic to the study drug or any of its auxiliary preparations;
* Patients with uncontrolled hypertension before enrollment, defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
* Patients with any disease or condition that affects drug absorption before enrollment, or patients who cannot take oral medication;
* Patients with active ulcers in the stomach and duodenum, ulcerative colitis or other digestive tract diseases before enrollment, or unremoved tumors with active bleeding, or other conditions that the investigator deems may cause gastrointestinal bleeding or perforation;
* Patients with obvious bleeding tendency evidence or history within 3 months before enrollment (bleeding > 30 mL within 3 months, accompanied by hematemesis, melena, or hematochezia), hemoptysis (fresh blood > 5 mL within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months;
* Patients with significant clinical cardiovascular diseases, including but not limited to acute myocardial infarction, severe/unstable angina or coronary artery bypass grafting within 6 months before enrollment; congestive heart failure with New York Heart Association (NYHA) classification > 2; drug-treated ventricular arrhythmias; left ventricular ejection fraction (LVEF) < 50%;
* Patients with active or uncontrolled severe infections (≥ CTCAE v5.0 grade 2 infections);
* Patients with known human immunodeficiency virus (HIV) infection. Patients with a history of clinically significant liver disease, including viral hepatitis [known hepatitis B virus (HBV) carriers must exclude active HBV infection, i.e., HBV DNA positive (> 1×104 copies/mL or > 2000 IU/mL); known hepatitis C virus (HCV) infection and HCV RNA positive (> 1×103 copies/mL)];
* Patients with any active autoimmune disease or a history of autoimmune disease (such as, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; patients with childhood asthma that has completely resolved and does not require any intervention in adulthood can be included; patients with asthma requiring medical intervention with bronchodilators cannot be included); replacement therapy is not considered systemic treatment, the following patients can be included: those with a history of autoimmune-related hypothyroidism and receiving thyroid hormone replacement therapy; type 1 diabetes that can be controlled with insulin treatment;
* Patients who have used immunosuppressants or systemic hormone therapy to achieve immunosuppression within 7 days before enrollment (dose > 10 mg/day of prednisone or other equivalent efficacy hormones);
* Patients with interstitial lung disease or pneumonia, pulmonary fibrosis, acute lung disease, or radiation pneumonitis;
* Pregnant (positive pregnancy test before medication) or lactating women; Any other disease, clinically significant metabolic abnormalities, physical examination abnormalities or laboratory test abnormalities, as judged by the investigator, there is reason to suspect that the patient has a disease or condition that is not suitable for the use of the study drug (such as having epilepsy and requiring treatment), or will affect the interpretation of the study results, or put the patient at high risk;
* Patients with urine routine indicating urine protein ≥ 2+ and 24-hour urine protein > 1.0g;
* Patients deemed unsuitable for inclusion in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | the duration from the date of randomization to any documented tumor progression or death due to any cause, assessed up to 12 months
  The rate of complete response and partial response

CONTACTS AND LOCATIONS:
Locations (1):
- Wanjing Feng, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We would like to share data if request.